CLINICAL TRIAL: NCT02736357
Title: The Lymphoma Epidemiology of Outcomes (LEO) Cohort Study
Acronym: LEO
Status: Withdrawn | Type: Observational
Why Stopped: Study restructured with Central IRB (NCT04996706); accruals reported there.
Sponsor: Mayo Clinic (Other)
Collaborators: Emory University (Other); University of Iowa (Other); M.D. Anderson Cancer Center (Other); Washington University School of Medicine (Other); University of Rochester (Other); Weill Medical College of Cornell University (Other); University of Miami (Other)
Responsible Party: Principal Investigator, James Cerhan, Principal Investigator, Mayo Clinic
Other Study IDs: 15-007282
Record Dates: First submitted 2016-04-04; First posted 2016-04-13 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: Lymphoma; Cohort; non-Hodgkin
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — Research blood draw collected at baseline. Research blood processed and stored as plasma, serum and germline DNA. Tissue in excess of diagnosis stored in formalin fixed paraffin embedded (FFPE) cored for use in Tissue Micro Array (TMA) and extraction of DNA and RNA from tumor.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this infrastructure grant is to establish and maintain a cohort of over 12,000 non-Hodgkin lymphoma (NHL) patients to support broad and cutting-edge research that identifies clinical (including co-morbid diseases), epidemiologic (including lifestyle and other exposures), host genetic, tumor, and treatment factors, as well as the interaction among these factors, on short and long-term outcomes. These efforts will identify new approaches to improve the survival and well-being of NHL patients.

DETAILED DESCRIPTION:
Newly diagnosed non-Hodgkin lymphoma (NHL) patients will be recruited from each center participating in the LEO cohort. At time of consent, participants will be asked to completed several questionnaires collecting health history, current medical and quality of life questions. Patients will also provide a baseline blood sample that will processed locally and stored centrally for future research use. Additionally, consent is given for use of excess clinical tumor tissue for research use.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed non-Hodgkin Lymphoma (NHL), within 183 days of enrollment
* Patients may have been treated as long as initial NHL diagnosis is within 6 months of enrollment
* 18 years of age or older

Exclusion Criteria:

* Lymphoma diagnosis greater than 184 days from date of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed non-Hodgkin Lymphoma willing to provide a research blood sample, return enrollment and follow-up questionnaires, and allow access to medical records.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-04-17 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | Short (<5 years), medium (5-10 years), and long-term (>10 years)
  Time from date of diagnosis to date of death

SECONDARY OUTCOMES:
Event Free Survival (EFS) | Short (<5 years), medium (5-10 years), and long-term (>10 years)
  Time from date of diagnosis to date of first defined event (disease progression, relapse or re-treatment for lymphoma, or death)
Lymphoma Specific Survival (LSS) | Short (<5 years), medium (5-10 years), and long-term (>10 years)
  Time from date of diagnosis to date of death due to lymphoma

CONTACTS AND LOCATIONS:
Overall Officials: James Cerhan, MD, PhD, Principal Investigator — Mayo Clinic; Christopher Flowers, MD, Principal Investigator — Emory University
Locations (8):
- United States (8):
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Weill Cornell Medical College, New York, New York
  - University of Rochester, Rochester, New York
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available.

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials